CLINICAL TRIAL: NCT05928117
Title: The Effect of Mobile Training Given in the Line of Coping With Fear of Birth on Fear of Birth, Birth Preference and Birth Experience
Brief Title: Training Given in the Line of Coping With Fear of Birth on Fear of Birth Birth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10.09.2021/49
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Birth; Fear of Childbirth; Education; Pregnancy; Fear
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Experimental and control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intervention: Mobile education given in the line of coping with fear The first one is 28-30th of pregnancy. week, the second is 36-38. It will meet in three meetings in total, the third of which will be within 12-24 hours postpartum.
  Interventions: Other: Education
- Control (No Intervention): Standart care

INTERVENTIONS:
Other: Education — Pregnant women will be given training to cope with the fear of childbirth.
  Other Names: Training to cope with the fear of childbirth education
  Arms: Experimental

SUMMARY:
Pregnancy and childbirth are a natural life event for women, as well as a process in which physical, biological and psychosocial changes are experienced. This process causes women to perceive childbirth as an unknown and unpredictable situation, resulting in the fear of childbirth. Due to the fear of childbirth, the daily routines, professional lives, social activities and relationships of pregnant women are significantly affected.

This study was planned to evaluate the effect of mobile education given in line with the "Guide to Coping with Fear of Birth" on fear of birth, birth preference and maternal satisfaction at birth. Research; It will be carried out at the T. C. Ministry of Health Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital. Data; The first one is 28-30th of pregnancy. week, the second is 36-38. It will meet in three meetings in total, the third of which will be within 12-24 hours postpartum. Data, Personal Information Form (Annex-1), Wijma Birth Expectation/Experience Scale (W-DEQ) Version A (Annex-2), Wijma Birth Expectation/Experience Scale Version B (Annex-3) and Birth Experience Scale ( Annex-4) and Postpartum Questionnaire (Annex-5). The obtained data will be analyzed with the SPSS 22.0 program.

In this study, it is thought that the training given to women with a high level of birth fear can reduce their fear of childbirth and increase maternal satisfaction at birth.

DETAILED DESCRIPTION:
The study is a randomized controlled management type study conducted to determine the effect of individual mobile training, which is reached by the "Guidelines for Coping with Fear of Birth" for primitive pregnant women.

Pregnancy and childbirth are a natural life event for women, as well as a process in which physical, biological and psychosocial changes are experienced. This process causes women to perceive childbirth as an unknown and unpredictable situation, resulting in the fear of childbirth. Due to the fear of childbirth, the daily routines, professional lives, social activities and relationships of pregnant women are significantly affected.

This study was planned to evaluate the effect of mobile education given in line with the "Guide to Coping with Fear of Birth" on fear of birth, birth preference and maternal satisfaction at birth. Research; It will be carried out at the T. C. Ministry of Health Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital. Data; The first one is 28-30th of pregnancy. week, the second is 36-38. It will meet in three meetings in total, the third of which will be within 12-24 hours postpartum. Data, Personal Information Form (Annex-1), Wijma Birth Expectation/Experience Scale (W-DEQ) Version A (Annex-2), Wijma Birth Expectation/Experience Scale Version B (Annex-3) and Birth Experience Scale ( Annex-4) and Postpartum Questionnaire (Annex-5).

ELIGIBILITY:
Inclusion Criteria:

* Primiparous,
* Having a single fetus,
* Able to read and write,
* Between the ages of 18-35,
* Volunteer to participate in the research,
* 28-30 days of pregnancy according to the last menstrual period or ultrasonography records. in the week,
* No risk factors (heart disease, placenta previa, oligohydramnios, preeclampsia, anhydramnios, diabetes, epilepsy),
* Having a telephone that can be contacted for mobile calls,
* Pregnant women who do not have any disability diagnosed for normal delivery.

Exclusion Criteria:

* Having communication problems,
* Having mental deficiency,
* Those who received infertility treatment and became pregnant with assisted reproductive techniques.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant
Enrollment: 67 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Fear of birth | Pre-test: Wijma Birth Fear/Experience version A and B were applied between 28-30 weeks of pregnancy. Post-test: Wijma Birth Fear/Experience version A and B were applied between 36-38 weeks.
  As the scale score increases, the fear of birth increases
Birth experience | Birth experience scale was applied between 12-24 hour
  As the score obtained from the scale increases, the mother has a good birth experience.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, PhD, Principal Investigator — Universty Of Cukurova
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No